CLINICAL TRIAL: NCT01159015
Title: A Multi-center, Double-masked, Randomized, Placebo-controlled, Parallel-group Study Evaluating the Safety of KetoNaph Ophthalmic Solution in Healthy, Normal Volunteers
Brief Title: Study Evaluating the Safety of KetoNaph Ophthalmic Solution in Healthy Volunteers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 586
Record Dates: First submitted 2010-07-06; First posted 2010-07-09 (Estimated); Results first posted 2020-09-14 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- KetoNaph (Experimental): KetoNaph Ophthalmic Solution
  Interventions: Drug: KetoNaph
- Vehicle (Placebo Comparator): Vehicle of KetoNaph Ophthalmic Solution
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: KetoNaph — Ophthalmic Solution administered BID for 6 weeks
  Arms: KetoNaph
Drug: Vehicle — Vehicle of KetoNaph ophthalmic solution administered bid for six weeks
  Arms: Vehicle

SUMMARY:
This study is being conducted to evaluate the safety of KetoNaph ophthalmic solution in healthy adult subjects and in pediatric subjects with a history or family history of ocular allergy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects less than 18 years of age, have either a history or family history of ocular allergy.
* ocular health within normal limits, including a calculated best-corrected visual acuity of 0.3 logMar or better, in each eye. For subjects under 10 years old who are developmentally unable to use the ETDRS chart, visual acuity will be made using the LEA symbols. For these subjects, 20-foot Snellen equivalent units of 20/63 or better in both eyes will be required.

Exclusion Criteria:

* Contraindications or sensitivities to the use of any of the investigational product(s) or their components.
* Subjects less than 18 years of age that have had symptoms and/or signs of allergic conjunctivitis/rhinitis and/or treatment with topical or systemic anti-allergy therapy, or have had a history of ragweed hypersensitivity during the 21-day period prior to visit 1.
* Surgical intervention within three months prior to Visit 1 or during the refractive surgery within the past 6 months.
* A known history of retinal detachment, diabetic retinopathy, or active retinal disease;
* An active ocular infection (bacterial, viral or fungal
* Use of any topical ophthalmic agents other than investigational products during study participation or within 5 days of beginning study treatment.
* Current or anticipated use of contact lenses during study participation or within 5 days of beginning study treatment.
* Current, prior (within 14 days of beginning study treatment) or anticipated use of systemic corticosteroids, and/or any other systemic medications which the Investigator feels may confound study data or interfere with the subject's study participation. Prior (within 21 days of beginning study treatment), current or anticipated use of any topical (including nasal) or systemic anti-allergy medications.
* Intraocular pressure (IOP) that is less than 5 mmHg or greater than 22 mmHg or have a normal IOP with a diagnosis of glaucoma.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tuyen Ong, MD, Principal Investigator — Bausch & Lomb Incorporated

RESULTS

PARTICIPANT FLOW:
Groups:
- KetoNaph: KetoNaph Ophthalmic Solution ketotifen fumarate 0.025%, naphazoline HCl 0.05%
  KetoNaph: Ophthalmic Solution administered BID for 6 weeks
Period: Overall Study
Arm/Group | KetoNaph | Vehicle
Started | 357 | 177
Completed | 339 | 170
Not Completed | 18 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KetoNaph | Vehicle | Total
Number analyzed (Participants) | 357 | 177 | 534
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.8 (17.2) | 31.0 (16.6) | 31.5 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 97 | 304
  Male | 150 | 80 | 230

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least One Adverse Event.
Description: An adverse event was defined as unfavorable and unintended sign, symptom, or disease temporally associated with the use of a test article, whether or not considered related to test article.
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | KetoNaph | Vehicle
Number analyzed (Participants) | 357 | 177
Participants | 113 | 34

ADVERSE EVENTS:
Time Frame: 42 days
Arm/Group | KetoNaph | Vehicle
Serious Adverse Events (participants affected / at risk) | 3/357 | 1/177
Other Adverse Events (participants affected / at risk) | 20/357 | 1/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KetoNaph (N=357) | Vehicle (N=177)
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Drug abuse (Psychiatric disorders) | 0 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KetoNaph (N=357) | Vehicle (N=177)
Eye Irritation (Eye disorders) | 20 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact sponsor directly for details.